CLINICAL TRIAL: NCT05650216
Title: A Single-arm，Single-center，Phase II Trial of Camrelizumab Combined With Neoadjuvant Concurrent Chemoradiotherapy for Resectable Locally Advanced Esophageal Squamous Cell Carcinoma（NICE-RT）
Brief Title: Camrelizumab Combined With Neoadjuvant Concurrent Chemoradiotherapy for Resectable Locally Advanced ESCC（NICE-RT）
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jun Liu, associate professor, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NICE-RT
Record Dates: First submitted 2022-11-24; First posted 2022-12-14 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Drug Therapy; Carboplatin; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunotherapy combined with Chemoradiotherapy (Experimental): A:Chemotherapy: nab-paclitaxel (80mg/m2), carboplatin (AUC=2)，on day 1,8,15,22,29;
  B:Immunotherapy: camrelizumab (200mg)，IV on days 5 and 26;
  C:Radiotherapy: Primary lesion and adjacent lymph nodes: 41.4Gy, 1.8Gy/23f; Abscopal lymph node 2Gy, 0.5Gy/4f.
  D:Ivor-Lewis or McKeown esophagectomy
  The participants will receive preoperative A+B+C. 4-6 weeks after completion of preoperative therapy ，D will be performed if there is no contraindication.
  Interventions: Drug: Chemotherapy (nab-paclitaxel AUC=2 and carboplatin 80mg/m2)，Immunotherapy (camrelizumab 200mg)、Radiotherapy(primary lesion and adjacent lymph nodes 41.4Gy， distant lymph node 0.5Gy*4)

INTERVENTIONS:
Drug: Chemotherapy (nab-paclitaxel AUC=2 and carboplatin 80mg/m2)，Immunotherapy (camrelizumab 200mg)、Radiotherapy(primary lesion and adjacent lymph nodes 41.4Gy， distant lymph node 0.5Gy*4) — 1. Neoadjuvant treatment period:
     Radiotherapy: Primary lesions and adjacent lymph nodes: The mode of involved field irradiation (IFI) is adopted, no preventive radiation is given. The total dose is 41.4Gy, 1.8Gy/23f. Distal lymph nodes ≥ 5cm away from the primary lesion: low-dose radiotherapy with a total dose of 4Gy, 0.5Gy/8f, Day1 to Day4, Day22 to Day25.
     Chemotherapy: Carboplatin(AUC=2), Nab-paclitaxel(80mg/m2), Day1/8/15/22/29. Immunotherapy: Camrelizumab(200mg, Day5, Day26).
  2. Perioperative period:
     Undergo surgery within 4-6 weeks after neoadjuvant therapy
  3. Adjuvant treatment period:
  Camrelizumab: (200mg, Q3W)，continued for up to 1 years，until PD or intolerable toxicity.
  Other Names: Camrelizumab: ai rui ka, SHR-1210; Nab-paclitaxel: ai yue

SUMMARY:
NICE-RT study is a "safety run-in" and phase II trial evaluating the safety and efficacy of Camrelizumab combined with Nab-paclitaxel and Carboplatin and Radiotherapy in patients with resectable locally advanced esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
Considering that immunotherapy combined with concurrent chemoradiotherapy may have unknown AEs, in order to explore the safety and tolerability of the regimen of camrelizumab combined with nab-paclitaxel and carboplatin and radiotherapy, this study set up an initial "safety run-in" phase. 10 patients will be firstly enrolled, and treatment-related adverse reactions（TRAEs）and surgical complications will be observed at the same time. If the completion rate of neoadjuvant therapy and surgery is greater than 80%, rate of 30-day major complication is less than 20%,and no death, it will continue to enroll 40 patients to explore the efficacy and safety of the regimen. If the completion rate of neoadjuvant therapy and surgery is less than 80%, the MDT will determine whether the study move forward. If treatment related death is more than 1 patients, the study will be terminated.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent has been signed.
2. In age from 18 to 75.
3. Thoracic esophageal squamous cell carcinoma confirmed by histology or cytology, which is classified as cT1b-4aN2-3M0 or M1 (only for supraclavicular lymph node metastasis), accompanied by lymph node metastasis (CT shows that the short diameter of the lymph node is greater than 1cm, the lymph node near the recurrent laryngeal nerve is greater than 8mm, the lymph node in the left upper abdominal region of the stomach is greater than 8mm, and PET-CT indicates positive).
4. At least one metastatic lymph node is more than or equal to 5cm from the primary lesion.
5. Have not received any anti-tumor treatment for esophageal cancer in the past, including radiotherapy, chemotherapy, surgery, etc.
6. The investigator assessed that lesion can be removed surgically.
7. At least one measurable lesion (according to RECIST 1.1)
8. ECOG PS: 0~1.
9. Weight loss<10% within 3 months, PG-SGA score<8.
10. Has sufficient organ function within 28 days before the first administration, (1) Blood routine: WBC≥3.0×109/L; ANC≥1.5×109/L; PLT≥50×109/L; HGB≥90 g/L (2) Liver function: AST≤5.0×ULN; ALT≤5.0×ULN; TBIL≤2.0×ULN (3) Renal function: Cr≤1.5×ULN or CrCl ≥60 mL/min (4) Coagulation function: INR≤1.5; APTT≤1.5×ULN (5)Women of childbearing age must take contraceptive measures within 3 months from the first dose to the last use of the study drug.

Exclusion Criteria:

1.Pathological type and stage

1. Pathology indicates that it is mixed squamous cell carcinoma (including adenosquamous carcinoma, squamous cell carcinoma, small cell carcinoma, carcinosarcoma, sarcomatoid carcinoma, etc.)
2. Non resectable or metastatic esophageal cancer

2. Medical history and complications

1. Subjects with any known active autoimmune disease (subjects who have stable clinical symptoms and do not need systematic use of immunosuppressants, such as type I diabetes and hypothyroidism that only need hormone treatment, and skin diseases that do not need systematic treatment can be included).
2. Subjects who have any complications requiring systemic treatment with glucocorticoids such as prednisone (>10mg/day) or who have used immunosuppressive drugs within 14 days before the first administration (subjects who do not have active autoimmune diseases, inhale or locally use glucocorticoids, and who use prednisone (>10mg/day) for hormone replacement treatment of adrenal insufficiency can be included in the group).
3. Subjects have received tumor vaccine or other immune activated anti-tumor drugs (such as interferon, interleukin, thymosin or immunocyte therapy) within 1 month before the first administration.
4. The subject is participating in other clinical trials or has received drug intervention from other clinical trials within 4 weeks before the first administration.
5. Subjects had received surgery or radiotherapy>30Gy within 4 weeks before the first administration.
6. Subjects with other malignant tumors that need to be treated (subjects with skin basal cell carcinoma, skin squamous cell carcinoma, breast cancer in situ or cervical cancer in situ that have received radical treatment and do not need other treatment can be included)
7. Subjects have suffered from serious cardiovascular diseases in the past: myocardial ischemia or myocardial infarction above Grade II, arrhythmia under poor control (including QTc interval ≥ 480 ms); Grade III-IV cardiac insufficiency; Color Doppler echocardiography showed that left ventricular ejection fraction (LVEF) was less than 50%.
8. Subjects have known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
9. Subjects received live vaccine within 30 days before the first administration.

3. Laboratory inspection

1. The subject's serum is HIV positive
2. Active hepatitis B (HbsAg positive and HBV-DNA ≥ 103 copies/mL) or active hepatitis C (HCV antibody positive and HCV-DNA positive, requiring antiviral treatment at the same time).

4. Allergies and adverse drug reactions should be excluded

1. Presence of allergy or hypersensitivity to monoclonal antibodies
2. Allergy or intolerance during infusion

5. Diseases or abnormal laboratory indicators that the investigator believes will affect the research results or are not in line with the interests of the subject should be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-12-25 (Estimated); Primary Completion 2023-12-25 (Estimated); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
Safety(The rates of grade 3 and higher-grade treatment-related adverse events) | From date of treatment allocation until surgery was applied during study period or up to at least 90 days after last dose
  Incidence of adverse events using CTCAE 4.03;grade 3 treatment-related adverse events and higher-grade adverse event will be reported
pCR | 12 months
  pathological complete response (pCR) is defined as disappearance of all invasive cancer after completion of neoadjuvant chemotherapy

SECONDARY OUTCOMES:
MPR | 12 months
  major pathologic response (MPR) is defined as residual viable tumor of less than or equal to 10%
ORR | 12 months
  objective response rate (ORR) is defined as the proportion of patients with a complete response(CR) or partial response(PR) to treatment according to RECIST v1.1
EFS | 12 months
  event-free survival (EFS) is defined as the time after treatment that a group of people in a clinical trial has not had cancer come back or get worse
OS | 12 months
  overall survival (OS) is defined as the time from treatment to death, regardless of disease recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Jun Liu, M.D., Principal Investigator — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China